CLINICAL TRIAL: NCT02040662
Title: Comparison of Continuous Epidural and Continuous Paravertebral Blockade in Postoperative Analgesia After Videothoracoscopic Lung Lobectomy
Brief Title: Comparison of Efficacy of Paravertebral and Epidural Analgesia After Videothoracoscopic Lung Lobectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmonary Hospital Zakopane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2014
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: paravertebral block; thoracic epidural analgesia; videothoracoscopic surgery; lung lobectomy
MeSH Terms: conditions — Lung Neoplasms | interventions — Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Thoracic Paravertebral Block (Experimental): 1. continuous thoracic paravertebral blockade 0,08 ml/kg/h with bupivacaine 0,25% + epinephrine 1:200.000
  2. patient-controlled analgesia (morphine), bolus dose 2 mg, lockout time 10 min
  Interventions: Procedure: Continuous Thoracic Paravertebral Block; Procedure: Patient-Controlled Analgesia with Morphine
- Continuous Thoracic Epidural Analgesia (Experimental): 1. continuous thoracic epidural block 0,06 ml/kg/h with bupivacaine 0,25% + epinephrine 1:200.000
  2. patient-controlled analgesia (morphine), bolus dose 2 mg, lockout time 10 min
  Interventions: Procedure: Continuous Thoracic Epidural Block; Procedure: Patient-Controlled Analgesia with Morphine

INTERVENTIONS:
Procedure: Continuous Thoracic Epidural Block — Before anesthesia, continuous thoracic epidural block of T5/T6 is performed (Portex Epidural Minipack set). Identification of paravertebral space by loss of resistance technique (air). A catheter is advanced ca. 3-5 cm, and test dose with 2 ml of lidocaine 2% i injected. At the end of surgery syringe with 0,25% bupivacaine with epinephrine 1:200.000 is connected to catheter and 6 ml bolus is injected, followed by an infusion of the same mixture at 0,06 ml/kg/h for postoperative pain management.
  Arms: Continuous Thoracic Epidural Analgesia
Procedure: Continuous Thoracic Paravertebral Block — Before anesthesia, continuous thoracic paravertebral block of T5/T6 is performed (Portex Epidural Minipack set). Identification of paravertebral space by loss of resistance technique (normal saline). After injection of 5-10 ml of normal saline a catheter is advanced medially ca. 5 cm. At the end of surgery syringe with 0,25% bupivacaine with epinephrine 1:200.000 is connected to catheter and 20 ml bolus is injected, followed by an infusion of the same mixture at 0,08 ml/kg/h for postoperative pain management
  Arms: Continuous Thoracic Paravertebral Block
Procedure: Patient-Controlled Analgesia with Morphine — Once arrived at the PACU all patients are placed on a postoperative analgesia regimen, that include:
  * patient-controlled analgesia with morphine (bolus dose 2 mg, lockout time 10 min)
  * paracetamol 1000 mg iv every 8 hrs
  * ketoprofen 100 mg iv every 12 hrs

SUMMARY:
Thoracic surgery correlates with significant pain in postoperative period. In order to alleviate the pain various combinations of pharmaceuticals and administration methods are employed. So as to reduce the extent of surgical trauma and, consequently, correlated pain various operation techniques are used. In traditional thoracotomy epidural anesthesia remains a golden standard. Epidural anesthesia however demands high skills to be performed correctly and presents an increased risk of grave complications. In videothoracoscopic (VATS) operations paravertebral blockade can be employed, yet there is no certainty if its efficacy after lung lobectomy. We therefore designed a prospective, randomized, parallel group, single site study to test the hypothesis, that continuous paravertebral blockade is as efficient in postoperative pain reduction as continuous epidural blockade and possesses a higher safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1-3
2. undergo videothoracoscopic lung lobectomy
3. forced expiratory volume in 1 second (FEV1) >1,5 l/min
4. no contraindications for epidural anesthesia and paravertebral nerve blockade
5. ability to comprehend principles of VAS pain examination method and to communicate in accordance with them.

Exclusion Criteria:

1. prior to the study: contraindications for local anesthesia, ASA>3, FEV1<1,5 l/min, conditions disabling the patient from comprehending the principles of VAS pain examination, known allergy to used medications.
2. during the study: failure to place epidural or paravertebral catheter, decision to abandon lobar resection (e.g. in case of neoplastic dissemination), intraoperative conversion to thoracotomy, intraoperative anatomical obstacles to distribution of local anesthetics, conditions disabling the patient from pain evaluation by means of VAS method (e.g. postoperative delirium), necessity to administer other pharmaceuticals influencing pain perception (e.g. sedatives), necessity of mechanical ventilation, interruption of local anesthesia as a result of technical problems (e.g. damage or slippage of catheter).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
pain intensity measured in VAS in predetermined time intervals after the operation | up to 96 hrs after the surgery

SECONDARY OUTCOMES:
respiratory parameters indirectly indicating conditions for efficient cough: peak expiratory flow (PEF), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) | up to 96 hrs after the surgery
frequency of side effects of regional anesthesia: urine retention resulting in necessity of bladder catheterization, hypotension, respiratory depression | up to 96 hrs after surgery
frequency of respiratory complications: atelectasis or pneumonia | up to 96 hrs after surgery
cumulative opioid (morphine) consumption | up to 96 hrs after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Hospital, Zakopane, Poland